CLINICAL TRIAL: NCT04300582
Title: Comparison Of The Fast Pharmaco-invasive Strategy With The Standard Pharmaco-invasive Strategy In Patients With ST Elevation Myocardial Infarction Stratified By The Forearm Approach: Randomized Clinical Trial
Brief Title: Fast Radial Pharmaco-invasive Strategy In ST Elevation Myocardial Infarction Trial
Acronym: FARADMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2020-01-06; First posted 2020-03-09 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2019-12

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
Keywords: stemi; thrombolysis; radial approach; acute coronary syndrome; pharmaco-invasive therapy; percutaneous coronary intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: Comparison of the fast pharmaco-invasive strategy with the standard pharmaco-invasive strategy in patients with ST-elevation myocardial infarction stratified by the forearm approach
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard pharmaco-invasive strategy (Active Comparator): Cardiac catheterization 3 to 24 hours after thrombolytic completion in STEMI patients.
  Interventions: Procedure: Cardiac catheterization standard strategy
- Fast pharmaco-invasive strategy (Experimental): Cardiac catheterization less than 3 hours after thrombolytic completion in STEMI patients.
  Interventions: Procedure: Cardiac catheterization fast strategy

INTERVENTIONS:
Procedure: Cardiac catheterization standard strategy — Cardiac catheterization by forearm approach 3 to 24 hours after thrombolytic completion in STEMI patients
  Arms: Standard pharmaco-invasive strategy
Procedure: Cardiac catheterization fast strategy — Cardiac catheterization by forearm approach within 3 hours after thrombolytic completion in STEMI patients
  Arms: Fast pharmaco-invasive strategy

SUMMARY:
INTRODUCTION: The pharmaco-invasive strategy is a safe alternative to primary percutaneous coronary intervention (PCI) in patients with ST elevation acute myocardial infarction, who cannot be in the cathlab in less than 120 minutes. However, previous studies of this strategy used the femoral artery as the main vascular access. Current studies show that the use of the radial artery in cases of acute myocardial infarction minimizes the risk of bleeding and mortality. Therefore, in the scenario where vascular access through the forearm vessels is recommended, the best timing to perform cardiac catheterization in the pharmaco-invasive strategy is not known.

OBJECTIVE: To compare the 24-hour hemoglobin drop (acute anemia) between the fast pharmaco-invasive strategy (within 3 hours) and the standard pharmaco-invasive strategy (3 to 24 hours) in patients with acute myocardial infarction (AMI) by coronary occlusion treated in Sancta Maggiore hospitals in São Paulo and underwent to cardiac catheterization through the forearm vessels.

METHOD: A prospective, randomized, multicenter study will be conducted in which 120 subjects will be randomly divided for fast and standard cardiac catheterization (1: 1). Stent implantation in the culprit vessel will be performed. The primary objective is to assess whether the fast cardiac catheterization is non-inferior to the standard strategy for a hemoglobin (Hb) drop within 24 hours. Considering in the control group an average drop of Hb 0.6 ± 1g / dl and that a drop greater than 3 g/dL of Hb is related to unfavorable clinical outcome, using a two-tailed alpha of 0.05 and a power of 90% to test the non-inferiority of the fast strategy with respect to standard strategy, each group will require 60 patients, totaling 120 individuals to include. However, if Hb fall in the fast strategy is greater than 3 g/dL and this result does not reproduce in the standard strategy, the study will allow us to show the superiority of the standard approach (between 3 and 24 hours).

DETAILED DESCRIPTION:
The FARAD MI will be a randomized, multicenter prospective study will be conducted. Patients with the diagnosis of ST-segment elevation acute myocardial infarction treated at the Sancta Maggiore Emergency Departments who have been thrombolyzed and aged up to 80 years will be included. After thrombolysis, patients will be immediately transferred to the Sancta Maggiore Hospital Itaim Unit and should arrive less than 3 hours after thrombolytic completion. When they arrive at the Interventional Cardiology Department, they will be explained about the study and offered to participate in the trial with consequent signature of the informed consent form. Thereafter, electrocardiogram and blood collection will be performed for laboratory tests, including hemoglobin, and patients will be randomized (1:1) to fast pharmaco-invasive strategy (within 3 hours of thrombolytic completion) and standard pharmaco-invasive strategy (3-24 hours). They will stay in the Interventional Cardiology Department until the procedure is performed and then the in-hospital care will be continued. Twenty-four hours after admission to the Interventional Cardiology Department, a new hemoglobin collection will be performed. Patients who refuse to participate in the trial will not have any harm in the treatment of acute coronary syndrome. Patients will receive standard clinical therapy, including dual antiplatelet therapy. Stent implantation will be performed in the culprit vessel by AMI. The treatment of residual coronary artery disease (coronary lesions with obstruction greater than 70% or with evidence of ischemia) will be discussed with the Clinical Cardiology team during hospitalization.

The following data will be collected: gender, age, ST-segment elevation location on the electrocardiogram (ECG), symptoms duration, time from first evaluation to ECG (door-to-ECG), time from first evaluation until thrombolytic administration (door-to-needle), thrombolytic used, medications administered at the origin unit, time between the end of thrombolytic and the beginning of cardiac catheterization, type of procedure (diagnosis and / or intervention), date and time of procedure, access site, radiation dose, contrast volume, associated comorbidities, laboratory, weight, height, BMI, coronary artery disease pattern (Syntax Score), vessel culprit for AMI, type and size of stent used, successful intervention, coronary flow at the end of the procedure (TIMI), angioplasty technique, residual coronary artery disease approach, bleeding (BARC), major cardiovascular adverse events (MACE), any cause and cardiovascular death. The hemoglobin of the patient's admission to the Interventional Cardiology Department and its variation after 24 hours will be evaluated. If red blood cell transfusion is required, pre-transfusion hemoglobin will be considered for evaluation.

Data from each patient will be registered in the REDCap platform in a electronic case report form (CRF) and will be submitted to statistical analysis using the Statistical Package for the Social Sciences (SPSS) 24 program. The REDCap has some important characteristics such as role-based authentication and security; real-time data validation and integrity checking; data assignment and audit capability; storage and sharing of protocols; central storage and backup of data and data export in formats compatible with known analysis programs as Excel, SPSS, Statistical Analysis System (SAS), Stata, R software, among others. Data will be audited by an independent team from Prevent Senior's Institute of Education and Research.

Patients who have the following characteristics will not be included in this trial: contraindications to fibrinolytic therapy, such as active internal bleeding, clinical signs of acute aortic dissection, traumatic or prolonged cardiopulmonary resuscitation (> 10 minutes), head trauma in the last four weeks, history of intracranial neoplasia, ischemic stroke in the past year or previous haemorrhagic stroke, pregnancy, sustained severe hypertension (≥180 mmHg systolic pressure and / or ≥110 mmHg diastolic pressure), trauma or major surgery in the last four weeks, use of oral anticoagulants, history of liver or kidney failure; did not meet reperfusion criteria upon arrival at the Interventional Cardiology Service of the Sancta Maggiore Hospital Itaim Unit (no improvement in chest pain or reduction in ST-segment elevation below 50% after thrombolytic administration); having femoral access as the first choice for invasive stratification; bleeding complications prior to cardiac catheterization, such as important hematoma and stroke; acute pulmonary edema (dyspnea of cardiac etiology with increased respiratory effort, hypoxemia and / or desaturation); cardiogenic shock (systolic blood pressure below 90 mmHg associated with signs of tissue hypoperfusion, such as oliguria, altered level of consciousness, cyanosis, cold and wet extremities, or vasopressor drug use); do not accept to sign the consent form.

Patients will be studied according to the precepts of the Helsinki Declaration and the Nuremberg Code, respecting the Research Norms Involving Human Beings (National Health Council resolution: 466/12) of the National Health Council. The study will be explained to patients when they are admitted to the Interventional Cardiology Department of the Sancta Maggiore Itaim Hospital and will be required to sign the Informed Consent Form (ICF) before any invasive procedure is performed. Randomization will be performed through a specific site after signing the consent form. The project was approved by the Research Ethics Committee of the Prevent Senior Research Institute.

To perform the sample calculation, the study of Bertrand OF et al (2010) was used to evaluate the variation of hemoglobin (Hb) in 24 hours after coronary angioplasty by radial approach. The control group had a mean hemoglobin drop of 0.6 ± 1g / dL and there were worse outcomes in patients with a hemoglobin drop greater than 3g / dL. (22) Therefore, considering in the control group a mean Hb fall of 0.6 ± 1g / dl and a fall greater than 3 g/dL of Hb is related to an unfavorable clinical outcome, using a two-tailed alpha of 0.05 and a power of 90% to test the non-inferiority of the fast strategy over the standard strategy, each group will require 60 patients, totaling 120 individuals to be included. However, if the Hb drop in the fast strategy is greater than 3 g/dL and this result does not reproduce in the standard strategy, the study will allow us to show the superiority of the strategy between 3 and 24 hours.

An intention-to-treat assessment will be performed. Categorical variables will be presented as absolute numbers and percentages. Continuous variables will be presented as mean ± standard deviation or median (interquartile range) according to their distribution. The distribution evaluation of continuous variables will be tested with Shapiro-Wilk. For continuous variables, the Student's t-test (normal distribution) or Wilcoxon-rank (non-normal distribution) will be used according to their distribution. For categorical variables the Chi-square test will be used.

ELIGIBILITY:
Inclusion Criteria:

* ST elevation myocardial infarction
* Submitted to thrombolysis
* Interventional Cardiology Department arrival less than 3 hours after the end of thrombolytic

Exclusion Criteria:

* Fibrinolytic therapy contraindication: active internal bleeding, clinical signs of acute aortic dissection, traumatic or prolonged cardiopulmonary resuscitation (> 10 minutes), head trauma in the last four weeks, history of intracranial neoplasia, ischemic stroke in the past year or previous haemorrhagic stroke, pregnancy, sustained severe hypertension (≥180 mmmHg systolic pressure and / or ≥110 mmHg diastolic pressure), trauma or major surgery in the last four weeks, use of oral anticoagulants, history of liver or kidney failure
* No reperfusion criteria when arriving at the Interventional Cardiology Department: no improvement in chest pain or reduction in ST-segment elevation below 50% after thrombolytic administration
* Femoral approach as the first choice for invasive stratification
* Bleeding complications before cardiac catheterization such as important hematoma and stroke
* Acute pulmonary edema: dyspnea of cardiac etiology with increased respiratory effort, hypoxemia and / or desaturation
* Cardiogenic shock: systolic blood pressure below 90 mmHg associated with signs of tissue hypoperfusion, such as oliguria, altered level of consciousness, cyanosis, cold and wet extremities, or vasopressor drug use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin change | 24 hours after cardiac catheterization
  Mean Hemoglobin change 24 hours after the cardiac catheterization

SECONDARY OUTCOMES:
Number of participants with Percutaneous Coronary Intervention failure | Immediately after percutaneous coronary intervention
  Patients with Final coronary minimum luminal diameter greater than 30% and / or final coronary flow TIMI 0 or 1 after percutaneous coronary intervention
Number of participants with net adverse clinical events (NACE) | Until hospital discharge, an average of 4 days
  Composite of death from all cause, and major bleeding (BARC 3 or 5) during hospitalization
Number of participants with hemoglobin change over 3 g/dL | 24 hours after cardiac catheterization
  Number of participants with hemoglobin change over 3 g/dL
Target vessel quantitative flow ratio (QFR) before the percutaneous coronary intervention | Immediately before the percutaneous coronary
  Target vessel quantitative flow ratio (QFR) before the percutaneous coronary intervention. This software measures the coronary flow after the procedure.
Target vessel quantitative flow ratio (QFR) after the percutaneous coronary intervention | Immediately after percutaneous coronary intervention
  Target vessel quantitative flow ratio (QFR) after the percutaneous coronary intervention. This software measures the coronary flow after the procedure.
Number of participants with ischemic or hemorrhagic stroke | Until hospital discharge, an average of 4 days
  Patients with ischemic or hemorrhagic stroke during hospitalization: loss of neurological function caused by an ischemic or hemorrhagic event with residual symptoms lasting at least 24 hours after onset or leading to death
All-cause death | Until hospital discharge, an average of 4 days
  All cause death during hospitalization
Number of participants with moderate bleeding: BARC 3a | Until hospital discharge, an average of 4 days
  Patients with overt bleeding plus hemoglobin drop of 3 to < 5 g/dL (provided hemoglobin drop is related to bleed); transfusion with overt bleeding
Number of participants with moderate bleeding: BARC 3b | Until hospital discharge, an average of 4 days
  Patients with overt bleeding plus hemoglobin drop > 5 g/dL (provided hemoglobin drop is related to bleed); cardiac tamponade; bleeding requiring surgical intervention for control; bleeding requiring IV vasoactive agents
Number of participants with moderate bleeding: BARC 3c | Until hospital discharge, an average of 4 days
  Patients with intracranial hemorrhage confirmed by autopsy, imaging, or lumbar puncture; intraocular bleed compromising vision
Number of participants with severe bleeding: BARC 5a | Until hospital discharge, an average of 4 days
  Patients probable fatal bleeding
Number of participants with severe bleeding: BARC 5b | Until hospital discharge, an average of 4 days
  Definite fatal bleeding (overt or autopsy or imaging confirmation)
Number of participants with reinfarction | Until hospital discharge, an average of 4 days
  New myocardial infarction during hospitalization: following the National Cardiovascular Data Registry (NCDR) criteria
Number of participants with recurrent angina | Until hospital discharge, an average of 4 days
  Recurrent angina during hospitalization: new angina after 6 hours of pci until discharge
Number of participants with heart failure | Until hospital discharge, an average of 4 days
  Number of participants with new or worsening heart failure during hospitalization: unusual dyspnea on light exertion, recurrent dyspnea occurring in the supine position, fluid retention; or the description of rales, jugular venous distension, pulmonary edema on physical exam, or pulmonary edema on chest x-ray
Number of participants with cardiogenic shock | Until hospital discharge, an average of 4 days
  Number of participants with cardiogenic shock during hospitalization: episode of systolic blood pressure <90 mm Hg, and/or cardiac index <2.2 L/min/m2 determined to be secondary to cardiac dysfunction for at least 30 minutes, and/or the requirement for parenteral inotropic or vasopressor agents or mechanical support (e.g., Intra aortic balloon pump (IABP), extracorporeal circulation, ventricular assist devices) to maintain blood pressure and cardiac index above those specified levels.
Number of participants with readmission | 30 days
  Number of participants with readmission after 30 days of index event
Number of participants with new revascularization of the target vessel | Until hospital discharge, an average of 4 days
  Number of participants with new revascularization of the target vessel during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Faillace, MD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Sancta Maggiore Hospital, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No